CLINICAL TRIAL: NCT00930046
Title: The Efficacy and Safety of Local Anesthetic Infusion With Ropivacaine for the Management of Pain After Surgical Correction of Ureteropelvic Junction Stenosis
Brief Title: The Efficacy and Safety of Local Anesthetic Infusion With Ropivacaine
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The institution transitioned from open surgical procedure to Robotic procedure
Sponsor: Boston Children's Hospital (Other)
Collaborators: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Principal Investigator, Navil Sethna, Senior Associate in Perioperative Anesthesia, Boston Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 08-11-0506
Record Dates: First submitted 2009-06-29; First posted 2009-06-30 (Estimated); Results first posted 2020-04-28 (Actual); Last update posted 2020-04-28 (Actual); Status verified 2020-02

CONDITIONS: Obstruction of Pelviureteric Junction
Keywords: ropivacaine; pediatric; children; continuous; wound; catheter; infusion; pyeloplasty
MeSH Terms: conditions — Multicystic renal dysplasia, bilateral; Wounds and Injuries

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ropivacaine group (Active Comparator): Patients in this group will receive ropivacaine via the wound catheter for the first 48hrs after surgery
  Interventions: Device: Ropivacaine wound catheter
- Normal Saline Group (Placebo Comparator): Will receive an infusion of normal saline for 48hrs post-operatively via the wound catheter.
  Interventions: Device: Saline wound catheter

INTERVENTIONS:
Device: Ropivacaine wound catheter — 19 gauge fenestrated wound catheter inserted into the fascial planes of the surgical site prior to skin closure with a separate exit site.
  Other Names: ON-Q Catheter
  Arms: Ropivacaine group
Device: Saline wound catheter — 19 gauge fenestrated wound catheter will be inserted into the fascial planes of the surgical site prior to wound closure
  Other Names: ON-Q Catheter
  Arms: Normal Saline Group

SUMMARY:
The investigators propose a prospective blinded randomized control trial (RCT) to assess the efficacy and safety of a simple method of continuous infusion of a local anesthetic, ropivacaine, via a surgical wound to control pain after ureteropelvic junction (UPJ) stenosis correction in children during the first 48 hrs after surgery. The investigators hypothesize that this technique will provide greater pain relief post-operatively and reduce the need for systemic opioid use along with a reduction in associated side effects of such analgesics.

DETAILED DESCRIPTION:
The investigators hypothesize that continuous infusion of local anesthetic via a wound catheter would improve postoperative pain control after UPJ correction and diminish the adverse effects associated with current use of opioids, administered via epidural or systemic route, for the management of postoperative pain. The expected benefits from wound catheter infusion are reduction in postoperative opioids requirement thereby diminishing the associated side effects of sedation, respiratory depression, nausea, vomiting, and ileus which occur at an average rate of 50% in children and adolescents based on recent meta-analysis. It may also facilitate early oral intake, ambulation and early discharge from the hospital.

The current use of epidural indwelling catheters for analgesia is associated with 20-25% technical failure rate from catheter misplacement, occlusion, disconnect or dislodgement, premature discontinuation of analgesia due to opioid-related side effects, requires bladder catheterization, and local anesthetic induced weakness in the lower extremities that usually delays ambulation. The dose of local anesthetics infused via the epidural route is much larger than proposed via wound catheters and carries greater risks of systemic toxicity compared to infusion doses anticipated via wound catheter infusion. In addition, the use of opioids such as morphine or hydromorphone via the epidural indwelling catheters produce adverse effects similar to that of systemic opioids and require electronic and close nursing monitoring.

Study Design

The study will include patients, male and female, between the ages of 3 months to 14 years of all ethnic and race groups. Patients with a history of clinically significant cardiovascular, pulmonary, hepatic, renal, neurologic, psychiatric or metabolic disease will be excluded. After obtaining consent from a legal guardian, patients will be randomly assigned to the placebo or treatment group. Both groups will receive rescue opioids for postoperative pain management via either patient-controlled analgesia (PCA) or nurse-controlled analgesia (NCA) administration for younger patients. The intraoperative anesthetic management will be standardized in all patients.

The wound catheter (Soaker multi-orifice catheter approved by the FDA) will be placed at the completion of the surgery in the subcutaneous space parallel and proximal to the surgical incision by the surgeon. The Pain Treatment Service will manage postoperative pain with standardized protocols including infusion of ropivacaine via the wound catheter and administration of rescue opioids via PCA/NCA. Patients will be randomly assigned to receive infusions of either ropivacaine or saline via the wound catheters.

Outcome Measures

The primary outcome measure is the total amount of opioids consumed by patients in the treatment group compared to that consumed by the placebo groups, noting the potential opioid-sparing effect in the patients treated with the continuous wound catheters with ropivacaine versus saline in the placebo group. The secondary outcome measures include a composite pain assessment scale (FLACC), that can be used as a self-report or observation scale, incidence of opioid-related incidence of nausea, vomiting, sedation and respiratory depression, time to first feed (as a measure of return of bowel function), transition to oral analgesics, time to first ambulation and time to discharge from the hospital. Finally, any adverse outcomes related to local anesthetic infusion, catheter related infection and technical failure such as catheter occlusion and premature dislodgement will be recorded.

Patient Recruitment

Patients will be identified from the Urology Clinic scheduling office and recruited in the Pre-operative Anesthesia Clinic.

Data Collection

Outcome measure data will be recorded by nurses and physicians who are unaware of the randomization for 48hrs post-operatively. The following outcome measures will be recorded. The total amount of opioids consumed by all patients over the first 48hrs after surgery, The daily total amount and pattern of opioid use via a PCA or NCA pump will be recorded from the electronic medical record. The pain assessment scores and adverse effects of opioids and local anesthetic administration will be recorded by a standardized protocol. Other outcome measures include the incidence of emesis, time to first feed or oral intake, pain intensity assessment by self-report in older children and observation in younger children, and time to discharge.

Statistical Analysis

Power analysis indicated that 48 patients randomized equally to each group (n=24 per group) will provide 80% (alpha= 0.05, beta= 0.20) power to detect a 25% difference in total opioid usage during the first 48 hours postoperatively. Fisher's exact test will be used to compare binomial proportions of nausea/vomiting, sedation, respiratory depression, ileus, and proportion of patients requiring postoperative opioids. In addition, groups will be compared using Kaplan-Meier curves and will be constructed to model time to first oral intake with the log-rank test to compare groups and 95% confidence intervals derived using Greenwood's formula. A Uniform(0,1) random number generator will be used to determine treatment allocation and to minimize any covariate imbalances between the ropivacaine and saline groups. Two-tailed values of p<0.05 will be regarded as statistically significant.

Summary

The investigators anticipate that the simple measure of wound catheter infusion with ropivacaine will demonstrate a significant safe and effective modality of analgesia in the postoperative period. If our results are valid, improved pain modulation with such a simple, low-tech modality of postoperative pain control (a) will require further investigation with a larger patient population including broader categories of surgical procedures to determine the limits of efficacy of such techniques in a particular surgical procedure, (b) may demonstrate statistically and clinically significant decreases in pain and decrease opioid demands, (c) may lessen time for recovery and side effects secondary to opioid use (d) offer significant cost-benefit for in-patient care relative to currently used modalities of epidural analgesia or systemic opioids for the management of postoperative pain in children undergoing UPJ correction and (e) compared to presently used epidural and PCA opioid analgesia, the wound catheter analgesia is expected to be less demanding on nurses and physicians (i.e. Pain Treatment Service), staff time, attention and need for close monitoring.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of UPJ stenosis requiring surgical repair
* Ages 3 months to 14 years old
* Guardians give consent and the child gives assent when appropriate
* Both genders
* All racial and ethnic groups

Exclusion Criteria:

* A history of chronic pain and/or use of chronic opioids and other analgesic(s)
* If parents/patients or attending urologist request epidural analgesia or refuse to participate in the study
* Impairment of cognition/neurologic, hepatic, renal, cardiovascular, endocrine, metabolic, and/or coagulation function
* A history of any diagnosis of psychiatric disorders, including bipolar disorders by self-report or by guardian
* A recent history of illicit chemical abuse within one week prior to surgical date
* Participants known to be taking prescribed medications or over-the-counter medications known to affect pain perception such as central nervous system stimulants, hypnotics, sedatives, etc within 24 hours of planned surgical procedure

Ages: 3 Months to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 15 (Actual)
Dates: Start 2009-04-24 (Actual); Primary Completion 2011-09-06 (Actual); Study Completion 2011-09-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Navil Sethna, MD, Principal Investigator — Boston Children's Hospital
Locations (2):
- United States (2):
  - Children's Hospital Boston, Boston, Massachusetts
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio

RESULTS

PARTICIPANT FLOW:
Groups:
- Ropivacaine Group: Patients in this group will receive ropivacaine via the wound catheter for the first 48hrs after surgery
  Wound catheter: 19 gauge fenestrated wound catheter inserted into the fascial planes of the surgical site prior to skin closure with a separate exit site.
- Normal Saline Group: Will receive an infusion of normal saline for 48hrs post-operatively via the wound catheter.
  wound catheter: 19 gauge fenestrated wound catheter will be inserted into the fascial planes of the surgical site prior to wound closure
Period: Overall Study
Arm/Group | Ropivacaine Group | Normal Saline Group
Started | 8 | 7
Completed | 7 | 5
Not Completed | 1 | 2
Not completed — Wound catheter malfunctioned | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ropivacaine Group | Normal Saline Group | Total
Number analyzed (Participants) | 8 | 7 | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 8 | 7 | 15
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 4 | 9
  Male | 3 | 3 | 6
Region of Enrollment [Number; unit: participants]
  United States | 8 | 7 | 15

OUTCOME MEASURES:

1. Primary Outcome: Morphine
Description: Total amount of morphine used in the first 48hrs immediately after surgery
Time Frame: 48 hours
Measure: Mean (Standard Deviation); unit: mg/kg per 48 hours
Arm/Group | Ropivacaine Group | Normal Saline Group
Number analyzed (Participants) | 7 | 5
mg/kg per 48 hours | 2.2 (1.8) | 3.5 (1.8)

2. Secondary Outcome: FLACC Pain Intensity [Faces Legs Activity Cry Consolability] 0-10 Points
Description: Observational FLACC pain intensity assessment tool that consists of observing the Faces Legs Activity Cry Consolability (FLACC) by the bedside nursing staff. This pain assessment tool is validated in non-verbal children and children at 7 years and younger.
  Minimum value is 0 and the maximum value is 10, where 0 represents no pain which is a better outcome.
Time Frame: 48 hours post-operatively
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Ropivacaine Group | Normal Saline Group
Number analyzed (Participants) | 7 | 5
score on a scale | 1.3 (0.7) | 1.9 (1.8)

ADVERSE EVENTS:
Time Frame: up to 48 hours post-operatively
Arm/Group | Ropivacaine Group | Normal Saline Group
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/7
Other Adverse Events (participants affected / at risk) | 0/8 | 0/7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No